CLINICAL TRIAL: NCT05615311
Title: Respiratory Outcomes After Early Vitamin D Supplementation in Infants Born Extremely Preterm: A Randomized Trial
Brief Title: Respiratory Outcomes After Early Vitamin D Supplementation in Infants Born Extremely Preterm
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ariel A. Salas, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 300010307
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prematurity; Extreme
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental)
  Interventions: Dietary Supplement: Vitamin D supplementation
- Control group (Placebo Comparator)
  Interventions: Other: No additional vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — Study participants assigned to the intervention group will receive 800 IU/ day of vitamin D plus 200-300 IU/day of vitamin D from parenteral and enteral sources during the first 2 weeks after birth.
  Arms: Vitamin D group
Other: No additional vitamin D supplementation — Study participants assigned to the control group will receive 200-300 IU/ day of vitamin D from parenteral and enteral sources during the first 2 weeks after birth.
  Arms: Control group

SUMMARY:
This is a masked randomized clinical trial in which extremely preterm infants fed human milk will be randomly assigned to receive either the highest (intervention group) or lowest (control group) vitamin D dose recommended during the first 14 days after birth.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 28 weeks or less

Exclusion Criteria:

* Major congenital anomalies and infants
* Terminal illness in whom decisions to withhold or limit life support have been made

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Severity of respiratory morbidity | 0 - 120 days
  A scoring system that defines severity of respiratory morbidity based on the amount of ventilatory support and the need for supplemental oxygen
Non-invasive oscillometry (NiOS) measurements of pulmonary mechanics | 40 - 120 days
  Using the tremoflo N-100 Neo Oscillometry device, we will determine the area under the reactance curve (AX)

SECONDARY OUTCOMES:
Bronchopulmonary dysplasia | 36 weeks PMA or discharge
  Number of participants receiving ventilatory support or supplemental oxygen at 36 weeks of postmenstrual age (PMA) or discharge

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Salas AA, Argent T, Jeffcoat S, Tucker M, Ashraf AP, Travers CP. Early Vitamin D Supplementation in Infants Born Extremely Preterm and Fed Human Milk: A Randomized Controlled Trial. J Pediatr. 2025 Dec;287:114754. doi: 10.1016/j.jpeds.2025.114754. Epub 2025 Jul 24. PMID 40714046